CLINICAL TRIAL: NCT00777374
Title: Single Center Phase I/IIa, Placebo Controlled, Randomized, Double-blind Preseasonal Study to Assess Clinical Efficacy and Safety of a Novel Method of Specific Allergen Immunotherapy in Grass Pollen Allergic Subjects by Epicutaneous Allergen Administration
Brief Title: Study of Specific Allergen Immunotherapy in Grass Pollen Allergic Subjects With Epicutanoeus Allergen Administration
Acronym: ZU-SkinSIT-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: PD Dr. Thomas Kündig, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZU-SkinSIT-003
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Allergic Rhinoconjunctivitis
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Allergen containing patch
  Interventions: Drug: Patch
- 2 (Placebo Comparator): Placebo patch
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Patch — epicutaneous application of allergen patch
  Arms: 1
Drug: Placebo patch — epicutanoeus application of a placebo patch
  Arms: 2

SUMMARY:
Seasonal rhinoconjunctivitis or hay fever is a common atopic condition that is frequently seen in clinical practice. Grass pollen is the major cause of pollinosis in many parts of the world. Immunotherapy is the only treatment that may affect the natural course of allergic diseases, and it may also prevent the development of asthma in patients with allergic rhinitis. With conventional subcutaneous desensitization the duration of treatment is around 3-5 years and usually comprises around 30-100 allergen injections. As high allergen doses have to be injected, allergic side effects may occur and patients must stay under medical supervision for at least 1 hour. Transcutaneous immunization (TCI) is a needle -free technique that delivers antigens and adjuvants to potent epicutaneous immune cells. The aim of the new epicutaneous route of desensitization is to more specifically target the immune system by loading Langerhans cells with the allergen. Lower antigen doses can be applied, such that side effects are reduced.

ELIGIBILITY:
Inclusion criteria: Written informed consent History of grass pollen allergic rhinitis for at least two years Male and female between 18 years to 65 years Positive skin-prick test to grass pollen Positive conjunctival provocation test

Exclusion criteria: Eczematous skin lesions on the upper arms Perennial rhinitis due to perennial allergies or anatomical reason (polyps, septal deviation) Symptoms of infectious disease with rhinitis in between the last week Surgical intervention in between the last 30 days Pregnancy or nursing History of HIV or AIDS History of mastocytosis (cutaneous or systemic) History of significant cardiovascular disease Uncontrolled Hypertension (blood pressure > 160 / 95) History of significant pulmonary, renal and/or hepatic disease History of significant hematological disorder Moderate or severe asthma History of malignancy Significant neurological or psychatric disease History of active autoimmune disease Antihistamines with longed half-lives in the last week Systemic or topical steroids for 5 days Depot corticosteroids for the last two months Active infectious disease Adipositas per magna

Contraindicated medications:

* immunosuppressive agents
* Betablockers
* ACE-inhibitors, AT 2 Antagonists
* tricyclic antidepressants
* daily use of Beta-agonists or steroid inhalers
* Participation in another clinical trial /study at the moment or within the last 60 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficacy of the placebo patch with the allergen patch with combined symptom medication score | 2009 - 2011

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland